CLINICAL TRIAL: NCT03781284
Title: Positron Emission Tomography With 18F-fluorodeoxyglucose Combined With MRI for Monitoring Inflammatory Activity in Patients With Ulcerative Colitis
Brief Title: PET Combined With MRI for Monitoring Inflammatory Activity in Patients With Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Crohn's and Colitis Foundation (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 360668
Record Dates: First submitted 2018-07-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Ulcerative Colitis
Keywords: [18F]-FDG PET/MR enterography; Diagnosis
MeSH Terms: conditions — Colitis, Ulcerative; Disease | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PET/MRI with bowel purgation (Experimental)
  Interventions: Diagnostic Test: [18F]-FDG PET/MRI; Diagnostic Test: Colonoscopy
- PET/MRI without bowel purgation (Experimental)
  Interventions: Diagnostic Test: [18F]-FDG PET/MRI; Diagnostic Test: Colonoscopy

INTERVENTIONS:
Diagnostic Test: [18F]-FDG PET/MRI
Diagnostic Test: Colonoscopy

SUMMARY:
Colonoscopy is considered crucial for the diagnosis and quantification of ulcerative colitis (UC). However, there are several drawbacks related to the invasiveness, procedure-related discomfort, risk of bowel perforation (especially in the period of acute inflammation), and relatively poor patient acceptance. Most patients regard the necessary bowel cleansing as burdensome. Feasible, accurate and well accepted non-invasive diagnostic techniques are needed for the determination of inflammatory activity and optimal tailoring of therapy. Hybrid PET/MRI represents an innovative combination of two established, non-invasive diagnostic tools: Magnetic resonance imaging (MRI), allowing for anatomic-functional imaging of the abdomen at high soft tissue contrast and positron emission tomography (PET) utilizing 18F-fluorodeoxyglucose (FDG) a non-invasive tool to monitor glucose metabolism and allowing a detection and quantification of inflammatory processes. Since MRI has limited sensitivity in UC and may be hampered by retained stool, a combination with another imaging modality is very appealing. PET, on the other side provides functional information, yet with limited anatomical landmarks and is relatively unsusceptible to artifacts associated to retained stool. In combination, these modalities might provide a valid alternative for the non-invasive assessment of the inflammatory activity in UC patients without the need for bowel purgation. It will therefore have to be investigated whether fecal material does impede the diagnostic quality of the combination of FDG-PET and MRI. For this purpose, the investigators will include 50 patients with confirmed ulcerative colitis. Dependent on clinical activity of the inflammation, patients will be randomized to undergo PET/MRI enterography either with or without prior bowel purgation followed by a colonoscopy. Inflammatory activity in 7 bowel segments will be analyzed based on PET/MRI with and without bowel purgation with the results of colonoscopy as standard of reference.

Patient acceptance of PET/MRI with and without bowel purgation as well as colonoscopy will be compared. PET/MRI with and without bowel cleansing will be compared with regard to diagnostic accuracy as well as for its patients' acceptance in comparison to colonoscopy.

The investigators hypothesize that PET/MRI will eventually be highly accurate to detect and monitor inflammatory activity in patients with ulcerative colitis. Additional information about extra-intestinal findings might also change the therapeutic concept. PET/MRI might serve as a non-invasive diagnostic option in patients with UC to quantify inflammatory activity especially when bowel cleansing or colonoscopy is not applicable.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed ulcerative colitis verified by the defining symptoms (rectal bleeding, diarrhea), endoscopy and histopathology
* clinically indicated colonoscopy and 18F-FDG PET as either initial assessment or follow- up examination
* patient age ≥ 18 years

Exclusion Criteria:

* Patients aged < 18years
* Patients with MRI contraindications, e.g. presence of cardiac pacemaker, implanted cardioverter-defibrillator, neurostimulation systems or with claustrophobia.
* acute renal failure, severe chronic renal failure (calculated glomerular filtration rate [GFR] < 30 ml/min)
* allergy to i.v. gadolinium based contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of PET/MRI with and without bowel purgation | 24 hours
  Overall segment-based diagnostic accuracy using ileocolonoscopy as reference standard will be calculated for PET/MRI with and without bowel purgation

SECONDARY OUTCOMES:
Sensitivity of PET/MRI with and without bowel purgation in percent | 24 hours
  Overall segment-based sensitivity using ileocolonoscopy as reference standard will be calculated for PET/MRI with and without bowel purgation
Specificity of PET/MRI with and without bowel purgation in percent | 24 hours
  Overall segment-based specificity using ileocolonoscopy as reference standard will be calculated for PET/MRI with and without bowel purgation
Negative predictive value of PET/MRI with and without bowel purgation in percent | 24 hours
  Overall segment-based negative predictive value using ileocolonoscopy as reference standard will be calculated for PET/MRI with and without bowel purgation
Positive predictive value of PET/MRI with and without bowel purgation in percent | 24 hours
  Overall segment-based positive predictive value using ileocolonoscopy as reference standard will be calculated for PET/MRI with and without bowel purgation
Optimized cut-offs | 24 hours
  Optimized cut-offs for PET for each bowel segment using ileocolonoscopy as reference standard for each colon segment will be calculated
Patient acceptance | 24 hours
  18F-FDG PET/MRI without bowel cleansing shows higher patient acceptance than conventional colonoscopy
Description of extraintestinal findings | 24 hours
  Extraintestinal findings will be assessed by evaluating PET/MRI images
The Boston Bowel Preparation Scale | 24 hours
  Bowel Preparation Quality will be assessed for both patient groups

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Khamou M, Schaarschmidt BM, Umutlu L, Forsting M, Demircioglu A, Haubold J, Koch AK, Bruckmann NM, Sawicki LM, Herrmann K, Boone JH, Langhorst J. Comparison of 18F-FDG PET-MR and fecal biomarkers in the assessment of disease activity in patients with ulcerative colitis. Br J Radiol. 2020 Aug;93(1112):20200167. doi: 10.1259/bjr.20200167. Epub 2020 Jun 24. PMID 32579403
- [Derived] Li Y, Schaarschmidt B, Umutlu L, Forsting M, Demircioglu A, Koch AK, Martin O, Herrmann K, Juette H, Tannapfel A, Langhorst J. 18F-FDG PET-MR enterography in predicting histological active disease using the Nancy index in ulcerative colitis: a randomized controlled trial. Eur J Nucl Med Mol Imaging. 2020 Apr;47(4):768-777. doi: 10.1007/s00259-019-04535-w. Epub 2019 Oct 24. PMID 31650217